CLINICAL TRIAL: NCT00813592
Title: A Phase II Study of SOM230 in Patients With Recurrent or Progressive Meningioma Who Have Previously Undergone or Are Not Candidates for Additional Surgery or Radiation
Brief Title: Phase II Study of SOM230 in Patients With Recurrent or Progressive Meningioma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Original PI left and company withdrew support.
Sponsor: University of Utah (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI26519
Record Dates: First submitted 2008-11-17; First posted 2008-12-23 (Estimated); Results first posted 2014-05-12 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Cancer
Keywords: meningioma; brain
MeSH Terms: conditions — Neoplasms; Meningioma | interventions — pasireotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All participants (Experimental)
  Interventions: Drug: SOM230B

INTERVENTIONS:
Drug: SOM230B — SOM230 is an injectable somatostatin analogue. Like natural somatostatin and other somatostatin analogues (SRIFa), SOM230 exerts its pharmacological activity via binding to somatostatin receptors (sst). There are five known somatostatin receptors: sst 1, 2, 3, 4 and 5. Somatostatin receptors are expressed in different tissues under normal physiological conditions. Somatostatin analogues activate these receptors with different potencies (Schmid and Schoeffter 2004) and this activation results in a reduced cellular activity and inhibition of hormone secretion. Somatostatin receptors are strongly expressed in many solid tumors, especially in neuroendocrine tumors where hormones are excessively secreted e.g. acromegaly (Freda 2002), GEP/NET tumors (Oberg, et al 2004) and Cushing's disease.
  Other Names: Pasireotide

SUMMARY:
This is a single-arm, phase II trial of SOM230 in patients with documented recurrent or progressive intracranial meningioma who have failed conventional therapy and are not candidates for complete surgical resection of their tumors and/or radiation at the time of study entry.

At the time of the final analysis, all patients who are receiving treatment with SOM230 will complete the core phase of the study and will continue on the extension phase. During this time, additional data on response duration, PFS, and safety will be collected.

DETAILED DESCRIPTION:
Study rationale/purpose:

Most, though not all (Lamberts 1995; Koper 1992) in vitro studies suggest that the addition of somatostatin inhibits meningioma growth, and accelerates apoptosis, suggesting a potential therapeutic role for somatostatin receptor agonists (Arena 2004). SOM230 (pasireotide) is a novel somatostatin analogue with affinity for multiple somatostatin receptors. Compared to octreotide (Sandostatin®), SOM230 binds to a wider spectrum of somatostatin receptors, including subtypes 1, 2, 3, and 5, and possesses as a higher binding affinity for subtypes 1, 3, and 5). In a recent study evaluating the expression of somatostatin receptor mRNA in human meningiomas (Arena 2004), 88% of the tumors (37/42) were positive for at least 1 of the 5 SSTR subtypes. SSTR1 and SSTR2 were most commonly detected in meningiomas (69 % (29/42) and 79% (33/42) respectively). The other subtypes were also frequently detected (43%, 33%, and 33% for SSTR3, SSTR4, and SSTR5 respectively). In recently completed studies with SOM230 in patients with Cushing's disease and acromegaly, clinical responses have been documented in patients who were refractory to Sandostatin. In summary, SOM230 has broader binding affinity to somatostatin receptors than Sandostatin®, its toxicity is very modest, and qualitatively identical to that of Sandostatin®, and its longer half-life (approximately 23 hours) allows a more convenient (twice daily in contrast to three times a day) dosing schedule compared with Sandostatin®. For all these reasons, we anticipate that the efficacy and tolerability of SOM230 in patients with recurrent meningiomas should be better than that observed with Sandostatin. We therefore, propose a formal phase II trial of SOM230 (pasireotide) in patients with recurrent or progressive meningiomas who have already undergone or are not candidates for additional surgery or radiation.

OBJECTIVES:

Primary objective To determine the objective response rate (ORR) (complete response [CR] plus partial response [PR]) of SOM230 monotherapy in patients with recurrent or progressive meningiomas who have previously undergone or are not candidates for additional surgery or radiation.

Secondary objectives

1. To determine the duration of response to SOM230
2. To establish the 6-month progression-free survival rate
3. To establish the median PFS and overall survival (OS)
4. To determine the clinical benefit rate (CR + PR + stable disease) of SOM230
5. To characterize the safety and tolerability of SOM230

Exploratory objectives

1. To determine the pharmacokinetic profile of SOM230
2. To analyze the expression of somatostatin receptor subtypes in tumor specimens (by immunohistochemistry) and in study participants (by octreotide scan). Please refer to sections 7.7.2 and 7.5.4.5 of the full protocol.
3. To measure serum IGF levels in patients prior to and after receiving SOM230
4. To determine the ORR for Grade 1 versus Grade 2 /3 meningiomas

SOM230 will be administered to all patients at a dose of 1200 µg given subcutaneously twice daily (Figure). One treatment cycle will be defined as four weeks of therapy. Complete blood counts will be obtained, and neurologic examinations and contrast-enhanced cranial MRI scans will be performed as described below (see Table 7-1). Serum IGF levels will be measured at the start of treatment, and at each MRI assessment point. Plasma pharmacokinetic studies will be performed in the subset of patients who consent to this additional study procedure. Participation in the pharmacokinetic component of this study is not mandatory.

All patients will continue to receive SOM230 until disease progression or death occurs, unacceptable toxicity is reported, or the patient declines further therapy.

In patients with stable (clinically unchanged or improved and radiographic disease increase or decrease in tumor size by less than 25%) or responding disease (clinically unchanged or improved and radiographic disease decrease in size by 50% or more), three additional cycles of SOM230 will be adminis¬tered, following which patients will be reassessed.

Post-Treatment Evaluation, Study Completion, and Survival Phase Study evaluation and determination of response status will be performed every 3 treatment cycles for the first 12 cycles of therapy and every 6 cycles thereafter for the duration of SOM230 treatment. At the time of the final primary analysis, all patients who are continuing to receive treatment with SOM230, as well as those who are being followed for post-treatment evaluations, and those who are being followed for survival only will complete the core phase of the study and will transition to the extension phase. During the extension phase, data on response duration, PFS and safety will continue to be collected.

Study completion will be declared following documentation of objective tumor progression by Macdonald and Levin criteria (either while on-treatment or during post-treatment evaluations) or at the time of death.

It is critical that objective tumor progression by Macdonald and Levin criteria be documented for each patient. In the event of treatment discontinuation prior to objective disease progression, patients will remain eligible for ongoing post-treatment evaluations. All antineoplastic therapies administered during the post-treatment phase will also be recorded as part of the post-treatment evaluation phase.

ELIGIBILITY:
PARTICIPANT SELECTION CRITERIA:

Inclusion Criteria:

1. Male or female patients aged 18 years or greater.
2. Patients with radiographically measurable disease and histologically confirmed recurrent or progressive intracranial meningiomas (refer to Appendix 1) who are not candidates for complete surgical resection of their tumors because the tumors are in eloquent areas of the brain (near critical neural structures)or are not candidates for cranial irradiation because a) they have already received radiation or b) the tumor is in close proximity to the optic nerve and radiation would likely result in vision damage.
3. Karnofsky Performance Status ≥ 60 (Requires occasional assistance, but is able to care for most of his/her personal needs.)
4. The following labs must not be clinically significant, as determined by PI. (Albumin, alkaline phosphatase, calcium, chloride, potassium, total protein, and sodium,)
5. Serum chemistries are as follows: bilirubin ≤ 1.5 X ULN, ALT or AST ≤ 2.5 X ULN, BUN ≤ 1.5X ULN, creatinine ≤ 1.5 X ULN.
6. Signed informed consent

Exclusion Criteria:

1. Patients receiving any cytotoxic chemotherapy, radiation or immunotherapy within 4 weeks prior to study enrollment
2. Patients who have undergone major surgery within 4 weeks(other than diagnostic surgery) or have not fully recovered, prior to study enrollment
3. Patients with malabsorption syndrome, short bowel syndrome, or chologenic diarrhea not controlled by specific therapeutic means
4. Patients with uncontrolled diabetes mellitus or a fasting plasma glucose > 1.5 ULN. Note: At the principle investigator's discretion, non-eligible patients can be re-screened after adequate medical therapy has been instituted.
5. Patients with symptomatic cholelithiasis
6. Patients who have congestive heart failure (NYHA Class III or IV), unstable angina, sustained ventricular tachycardia, ventricular fibrillation, clinically significant bradycardia, advanced heart block, or a history of acute myocardial infarction within the six months preceding enrollment.
7. Patients with congenital QTc syndrome, drug-induced prolonged QTc interval, or QTc measurement > 450 msec.
8. Patients with liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis with serum bilirubin > 1.5 X ULN, and/ or ALT or AST > 2.5 X ULN
9. Patients with prior or concurrent malignancy except for the following: adequately treated basal cell or squamous cell skin cancer, or other adequately treated in situ cancer, or any other cancer from which the patient has been disease free for five years.
10. Patients with active or suspected acute or chronic uncontrolled infection or with a history of immunocompromise, including a positive HIV test result (ELISA and Western blot).
11. Patients with ANC <1.5 X 109/L; Hgb <10 g/dL; PLT <100 X 109/L
12. Patients who have any current or prior medical condition that, in the opinion of the Investigator, may interfere with the conduct of the study, the evaluation of its results, or the rigorous completion of the informed consent process.
13. Female patients who are pregnant or lactating, or adults of childbearing potential who are not practicing a medically acceptable method of birth control. Female patients must use barrier contraception in addition to condom use in their partner. If oral contraception is used, the patient must have been practicing this method for at least two months prior to enrollment and must agree to continue the oral contraceptive throughout the course of the study, and for three months after the study has ended. Male patients who are sexually active are required to use condoms during the study and for three months afterward.
14. Patients who have participated in any clinical investigation with an investigational drug (other than SOM230) within 1 month prior to study drug dosing.
15. Known hypersensitivity to somatostatin analogues or any component of the pasireotide or octreotide LAR or s.c. formulations (see section 6.1.1)
16. Patients with a history of non-adherence to medical regimens or who are considered potentially unreliable or will be unable to complete the entire study
17. QTcF at screening > 450 msec.
18. History of syncope or family history of idiopathic sudden death.
19. Sustained or clinically significant cardiac arrhythmias.
20. Risk factors for Torsades de Pointes such as hypokalemia, hypomagnesemia, cardiac failure, clinically significant/symptomatic bradycardia, or high-grade AV block.
21. Concomitant disease (s) that could prolong QT such as autonomic neuropathy (caused by diabetes, or Parkinson's disease), HIV, cirrhosis, uncontrolled hypothyroidism or cardiac failure.
22. Concomitant medication (s) known to increase the QT interval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randy Jensen, MD, Principal Investigator — University of Utah
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: SOM230B : SOM230 is an injectable somatostatin analogue. Like natural somatostatin and other somatostatin analogues (SRIFa), SOM230 exerts its pharmacological activity via binding to somatostatin receptors (sst). There are five known somatostatin receptors: sst 1, 2, 3, 4 and 5. Somatostatin receptors are expressed in different tissues under normal physiological conditions. Somatostatin analogues activate these receptors with different potencies (Schmid and Schoeffter 2004) and this activation results in a reduced cellular activity and inhibition of hormone secretion. Somatostatin receptors are strongly expressed in many solid tumors, especially in neuroendocrine tumors where hormones are excessively secreted e.g. acromegaly (Freda 2002), GEP/NET tumors (Oberg, et al 2004) and Cushing's disease.
Period: Overall Study
Arm/Group | All Participants
Started | 2
Treated | 2 (Two patients were treated.)
Response Assessment | 1 (One patient met the response assessment.)
Completed | 0
Not Completed | 2
Not completed — Disease assessment was not completed per | 2

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) of SOM230 Monotherapy in Meningioma
Description: Measured the percentage of participants achieving a complete response or partial response as opposed to those participants with progressive disease or stable disease.
Time Frame: November 2011
Arm/Group | All Participants
Number analyzed (Participants) | 0

2. Secondary Outcome: To Determine the Duration of Response to SOM230
Time Frame: November 2011
Arm/Group | All Participants
Number analyzed (Participants) | 0

3. Secondary Outcome: To Establish the 6-month Progression-free Survival Rate
Time Frame: November 2011
Arm/Group | All Participants
Number analyzed (Participants) | 0

4. Secondary Outcome: To Establish the Median PFS and Overall Survival (OS)
Time Frame: November 2011
Arm/Group | All Participants
Number analyzed (Participants) | 0

5. Secondary Outcome: To Determine the Clinical Benefit Rate (CR + PR + Stable Disease) of SOM230
Time Frame: November 2011
Arm/Group | All Participants
Number analyzed (Participants) | 0

6. Secondary Outcome: To Characterize the Safety and Tolerability of SOM230
Description: Number of participants to experience adverse events
Time Frame: Monthly from study entry until subject taken off study, average 28 months
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 2
participants | 2

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=2)
elevated glucose level (Blood and lymphatic system disorders) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
foot pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes